CLINICAL TRIAL: NCT02901652
Title: Comparison of Nasal Intermittent Positive Airway Pressure and Nasal Bi-level Positive Airway Pressure Methods in Preterm Infants With Respiratory Distress Syndrome With Gestational Age of 26-30 Weeks
Brief Title: NIPPV and nBiPAP Methods in Preterm Infants With Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02082016
Record Dates: First submitted 2016-08-02; First posted 2016-09-15 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2018-10

CONDITIONS: Prematurity; Respiratory Distress Syndrome
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIPPV (Active Comparator): noninvasive respiratory support devices
  This group receiving Nasal Intermittent Positive Pressure Ventilation (NIPPV) treatment.
  Interventions: Device: noninvasive respiratory support devices
- BİPAP (Active Comparator): noninvasive respiratory support devices
  This group receive Bi-Level Positive Airway Pressure (BIPAP) treatment.
  Interventions: Device: noninvasive respiratory support devices

INTERVENTIONS:
Device: noninvasive respiratory support devices

SUMMARY:
Purpose is to compare introduction of NIPPV (Nasal Intermittent Positive-Pressure Ventilation) and nBiPAP (Nasal Bi-level Positive Airway Pressure) in terms of mechanical ventilation (MV) need (non-invasive respiratory support failure) and surfactant need within the first 72 hours of life in preterm infants with Respiratory Distress Syndrome (RDS) at 26-30 weeks of gestation.

DETAILED DESCRIPTION:
Purpose is to compare introduction of NIPPV and nBiPAP in terms of mechanical ventilation (MV) need (non-invasive respiratory support failure) and surfactant need within the first 72 hours of life in preterm infants with Respiratory Distress Syndrome (RDS) at 26-30 weeks of gestation.

Method

Primary Outcome Measures:

In NIPPV and BIPAP groups, comparison of mechanical ventilation (MV) need (non-invasive respiratory support failure) and surfactant need within the first 72 hours of life

Secondary Outcome Measures:

* Compare patients' need of total duration of invasive and non-invasive respiratory support and the duration of free oxygen
* Compare oxygen need in postnatal day 28 and week 36
* Compare the presence and severity of BPD (Bronchopulmonary dysplasia)
* Compare premature morbidities such as PDA (patent ductus arteriosus), IVH (intraventricular haemorrhage), NEC (necrotizing enterocolitis), ROP (retinopathy of prematurity)
* Compare feeding intolerance, reaching birth weight and transition to full oral feeding time, hospitalization period
* Compare their neurodevelopment in postnatal age 2

Study Design In NIPPV group; non-synchronous mode will be used, and they will be titrated between FiO2: 021-0.50 in a respiratory rate of 20-40 / min, peak inspiratory pressure (PIP): 15-20 end-expiratory pressure (PEEP):5-6 cm H2O and target oxygen saturation: 90-95 %. In nBiPAP group; they will be titrated between 021-0.50, in non-synchronized PEEP:6 H2O, pressure amplitude: 3 cm H2O, FiO2 target oxygen saturation of 90-95 %.

Under non-invasive respiratory support, in case of FiO2 is ≥ 0.40, surfactant will be given as early rescue therapy by means of non-invasive method (by using a thin catheter - take care method- while spontaneous breathing continues) in order to keep target oxygen saturation between 90-95 %. The second dose of surfactant will be given 6 hours after the first dose by means on non-invasive method in order to keep target oxygen saturation between 90-95 % in case of FiO2 need is ≥ 0.30.

Non-invasive respiratory support failure is set as follows:

* FiO2 of ≥ 0.50 in order to keep oxygen saturation measured by pulse oximetry above 90 % and higher,
* Apnea requiring more than 6 alerts in a 24 -hour period in 6 consecutive hours or more than 1 apnea requiring positive pressure ventilation,
* Persistent acidosis; presence of pH < 7.20 and PCO2 > 65 mmHg in two different blood gases drawn with an interval of at least 30 minutes or treatment-resistant metabolic acidosis,
* Severe respiratory distress,
* Pulmonary haemorrhage and cardiopulmonary arrest.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant with gestational age of 26 weeks 0 days and 29 weeks 6 days will be included.

Exclusion Criteria:

* Major congenital anomalies
* Presence of cardiovascular instability
* Intubation at admission to the NICU
* Consent not provided or refused

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 325 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
surfactant requirement | 72 HOURS
  surfactant requirement within the first 72 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Suna Oğuz, MD, Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching, Ankara, Turkey (Türkiye)